CLINICAL TRIAL: NCT00691899
Title: A Phase III Study to Assess the Safety, Tolerability, and Efficacy of MK0822 (Odanacatib) in Prolonging Time to First Bone Metastasis in Men With Castration-Resistant Prostate Cancer
Brief Title: A Study to Assess the Effects of MK0822 in Prolonging Time to First Bone Metastasis in Men With Castration-Resistant Prostate Cancer (0822-030)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn for administrative reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0822-030; 2006_533; MK-0822-030
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: odanacatib
- 2 (Placebo Comparator)
  Interventions: Drug: placebo (unspecified)

INTERVENTIONS:
Drug: odanacatib — odanacatib; 5mg oral, once daily for Approximately 36 months.
  Other Names: MK0822
  Arms: 1
Drug: placebo (unspecified) — placebo; oral, once daily for Approximately 36 months
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effects of MK0822 in prolonging the time to first bone metastasis in men with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Merck Duration of Treatment : odanacatib; approximately 36 months (even driven study) - Comparator Duration of Treatment : placebo (unspecified); approximately 36 months (event driven study)

ELIGIBILITY:
Inclusion Criteria:

* Castration-resistant prostate cancer; increased risk for prostate cancer progression
* Patient underwent bilateral orchiectomy 6 months or more (i.e., =180 days) prior to Visit 1, or is receiving androgen-deprivation therapy and is on a stable regimen for at least 3 months (i.e., =90 days) prior to Visit 1. Androgen-deprivation therapy may include gonadotropin-releasing hormone agonists such as leuprolide, goserelin, or triptorelin

Exclusion Criteria:

* Bone metastases or history of bone metastases
* Patient has other distant metastases (e.g., visceral, including brain, or soft-tissue). Patients with regional lymph nodal metastases are eligible
* Patient has ANY of the following:

  1. currently is receiving a bisphosphonate or other drug therapy for osteoporosis
  2. has been treated with an oral bisphosphonate for osteoporosis for more than 3 months within the 2 years prior to Visit 1, or for a total of more than 6 months at any time prior to Visit 1
  3. has been treated with an intravenous bisphosphonate within the 12 months prior to Visit 1
* Patient has received chemotherapy within the 2 years prior to Visit 1 (for example, doxorubicin, cytoxan, estramustine, paclitaxel, docetaxel, etoposide, vinblastine, 5-fluorouracil, interferon, mitoxantrone). This exclusion criterion does not include androgen-deprivation therapy (e.g., gonadotropin-releasing hormone agonists such as leuprolide, goserelin, or triptorelin)
* Patient has a history of any malignancy other than prostate cancer <5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer. Melanoma, leukemia, lymphoma, and myeloproliferative disorders of any duration are excluded
* Patient is currently participating in, or has participated in a study with an investigational compound or device within 30 days of signing the informed consent
* Patient is currently participating in or has at any time in the past participated in a prostate cancer study with a registered medication (i.e., approved by the regulatory agency in which he resides) being tested for the treatment of prostate cancer (an unapproved indication)
* Patient is currently using a systemically administered azole antifungal (for example, ketoconazole, fluconazole, itraconazole, miconazole, posaconazole, ravuconazole, and voriconazole). Patients taking these medications must discontinue their use at least one week prior to starting blinded study medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of treatment with MK0822 5 mg once daily on bone metastasis-free survival (i.e., the risk of developing a first bone metastasis or dying from any cause) compared to placebo | Approximately 36 months (event-driven study)

SECONDARY OUTCOMES:
To assess the effect of treatment with MK0822 5 mg once daily on the risk of developing a first bone metastasis compared to placebo | Approximately 36 months (event-driven study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC